CLINICAL TRIAL: NCT00808327
Title: Spinal Anesthesia for Cesarean Delivery: Bupivacaine With or Without Fentanyl
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Dr. Alison Macarthur, Mount Sinai Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 08-03
Record Dates: First submitted 2008-12-11; First posted 2008-12-15 (Estimated); Last update posted 2009-11-20 (Estimated); Status verified 2009-11

CONDITIONS: Pain
Keywords: Cesarean section; Spinal
MeSH Terms: conditions — Pain | interventions — Bupivacaine; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Bupivacaine alone
  Interventions: Drug: Bupivacaine
- 2 (Active Comparator): Bupivacaine plus Fentanyl
  Interventions: Drug: Bupivacaine, fentanyl

INTERVENTIONS:
Drug: Bupivacaine — A single, 15mg, intrathecal dose of bupivacaine.
  Other Names: Marcaine
  Arms: 1
Drug: Bupivacaine, fentanyl — A single, 12 mg, intrathecal dose of bupivacaine, plus 15 micrograms of fentanyl
  Other Names: Marcaine
  Arms: 2

SUMMARY:
The safest form of anesthesia for Cesarean section is a spinal anesthetic. All spinal anesthetics contain a local anesthetic and/or a narcotic. A drug named bupivacaine is the most commonly used local anesthetic in spinal anesthetics for Cesarean deliveries in North America. Another drug named fentanyl is the most commonly used narcotic. This study will look at whether a spinal anesthetic with 15mg of bupivacaine alone will be the same as a spinal anesthetic with 12mg of bupivacaine and 15ug of fentanyl.

DETAILED DESCRIPTION:
There have been many studies looking at different doses and combinations of bupivacaine and fentanyl but there is no agreement among anesthesiologists as to the best combination of drugs.

The main problem with bupivacaine is that it causes hypotension (low blood pressure). When fentanyl is added to bupivacaine, a lower dose of bupivacaine can be used so that there is less of a fall in blood pressure. The main problem with fentanyl is itchiness and sleepiness. In the case of an emergency Cesarean section, the extra time needed to draw-up and administer a second medication may make a difference to the health of the baby.

Our goal is to determine whether high dose bupivacaine (15mg) alone will produce spinal anaesthesia for cesarean delivery equivalent to 12mg of intrathecal hyperbaric bupivacaine in combination with 15ug of intrathecal fentanyl.

ELIGIBILITY:
Inclusion Criteria:

* healthy patients (ASA 1 or 2)
* BMI < 40
* height between 5 & 6 feet

Exclusion Criteria:

* parturients with pregnancy induced hypertension or preeclampsia
* parturients with significant cardiac, renal or other organ-system disease which preclude choice of spinal anesthesia
* emergency delivery
* triplet or greater multiple gestation

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 140 (Actual)
Dates: Start 2009-01; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
The primary outcome is the maximal degree of abdominal sensation felt by the patient during surgery. | 1 hour

SECONDARY OUTCOMES:
Speed of onset of block to T4 dermatome (minutes), as well as highest level of block (dermatomal level) and degree of motor block (Bromage scale) | 30 minutes
The degree of patient discomfort will be evaluated using a 10 cm linear visual analog scale (VAS). | 1 hour
The amount of additional IV analgesia administered during the intraoperative period. | 1 hour
Time to regression of block (minutes) | 4 hours
Duration of analgesia (hours) | 24 hours
Incidence of side effects: Intraoperative pruritus, nausea and vomiting in the absence of hypotension, somnolence, shivering, euphoria or dysphoria and respiratory depression will be evaluated. | 2 hours
Dose of vasopressor(s) given during surgery | 1 hour
Lowest Mean Arterial Pressure during surgery (=2/3 diastolic pressure + 1/3 systolic pressure). | 1 hour
Patient satisfaction. A number of questions answered on a Likert Scale will be asked post-Cesarean section. | 15 minutes
Neonatal arterial blood gas results (pH) and 1 and 5-minute APGAR scores (1 - 10) will be recorded | 10 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Alison J Macarthur, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada